CLINICAL TRIAL: NCT05561556
Title: Mitochondria Dysfunction as a Contributor to Racial Disparities in Vascular Health and Hypertension
Brief Title: Mitochondria Oxidative Stress and Vascular Health Study
Acronym: MOVHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Austin Robinson, Assistant Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AU IRB #22-154
Record Dates: First submitted 2022-09-15; First posted 2022-09-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases; Hypertension; Racism; Vascular Diseases
Keywords: Cardiovascular health; Hypertension; Health disparities; Renal function; Vascular health
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Racism; Vascular Diseases | interventions — mitoquinone

STUDY DESIGN:
Intervention Model Description: The intervention is to give participants an 8-week supplementation of one capsule (20 mg) of either a mitochondrial antioxidant (MitoQ) or a placebo (dextrin and silica), in a randomized order. Followed by a two-week washout, then another 8-week supplementation of a 20 mg capsule.
Who Masked: Outcomes Assessor
Masking Description: The member of the study team performing data analysis will be blinded when performing data analysis and unblinded after the final statistical analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitoQ (Experimental): 8-week MitoQ supplementation (20 mg daily capsule).
  Interventions: Dietary Supplement: MitoQ
- Placebo (Placebo Comparator): 8-week placebo matched in appearance to MitoQ supplementation (20 mg daily capsule).
  Interventions: Dietary Supplement: MitoQ

INTERVENTIONS:
Dietary Supplement: MitoQ — One 20mg capsule daily for 8 weeks

SUMMARY:
Cardiovascular diseases (CVDs) are the number one cause of death in America and most of the post-industrial world. Hypertension is a leading risk factor for CVDs including stroke, myocardial infarction, and heart failure. Black Americans suffer from the highest rates of hypertension of any racial/ethnic group in America, among the highest in the world. There are also well-documented racial disparities in vascular dysfunction (e.g., endothelial dysfunction, arterial stiffening). Thus, racial disparities in hypertension and vascular dysfunction exacerbate the burden of CVDs, with Black Americans being 30% more likely to die from CVD than any other race in the US. It is established that mitochondrial dysfunction contributes to vascular dysfunction. However, there is a knowledge gap regarding whether targeting mitochondrial dysfunction attenuates oxidative stress, vascular dysfunction, and CVD risk among Black adults at heightened CVD risk. Thus, the investigators will conduct an 8-week trial with the mitochondrial antioxidant MitoQ in middle-aged and older Black and non-Black adults. Our overarching hypothesis is that mitochondrial dysfunction contributes to heightened oxidative stress, vascular dysfunction, and higher BP in Black adults; and that MitoQ will attenuate these racial differences. Importantly, the investigators will also assess social determinants of health (e.g., income, neighborhood disadvantage, discrimination) and health behaviors (e.g., diet, physical activity) and uncover their role in oxidative stress, vascular function, and BP Regarding methodology, the investigators will perform blood draws, vascular testing, preceding and following an 8-week, 20mg daily consumption of MitoQ and placebo. The investigators will also measure urine biomarkers of kidney function and blood pressure in adults (45-75 years old).

DETAILED DESCRIPTION:
Hypertension develops earlier in life, is more challenging to control, and is associated with greater rates of morbidity, such as end-organ damage (e.g., kidneys) in Black compared to White adults. Recently published data from the Coronary Artery Risk Development in Young Adults (CARDIA) study5 demonstrate that the cumulative incidence of hypertension by age 55 was 76% in Black adults (both males and females), 55% in White males, and 40% in White females and that racial differences in blood pressure (BP) started to emerge as early as the third decade of life. Data from Bogalusa Heart Study suggest that Black individuals have higher BP levels as early as childhood. Black Americans' hypertension rates exceed any other race/ethnic group (not just non-Hispanic White) in America. Black Americans also tend to have worse BP than foreign-born Black adults, indicating a role of socioeconomic factors. The AHA has projected that between 2010 and 2030, direct medical costs of cardiovascular diseases (CVDs) are projected to triple, from $273 billion to $818 billion. Moreover, recent projections demonstrate that the annual costs of health disparities in preventable chronic diseases will increase to $50.1 billion by 2050. Given the alarming public health and economic consequences of hypertension and CVDs, addressing the issue of racial disparities in hypertension to reduce the burden of CVDs is critical. A key contributor to disparities in hypertension and CVD is vascular dysfunction. Several studies have demonstrated racial disparities in endothelial function, arterial stiffness, and autonomic control of BP including exaggerated BP responses to sympathoexcitatory stimuli, such as exercise. However, the underlying mechanisms for the racial difference in vascular dysfunction are still unknown. Excess oxidative stress (i.e., ROS) contributes to racial differences in endothelial function. Black males exhibit greater resting PBMC-derived ROS production which could contribute to increased systemic oxidative stress. Multiple publications also demonstrate that excess ROS contributes to microvascular dysfunction in young non-Hispanic Black compared to non-Hispanic White adults. NADPH oxidase and xanthine oxidase inhibition did not fully attenuate the racial disparity in microvascular function, suggesting that an alternative source of ROS, such as the mitochondria, may play a role in racial disparities in endothelial function. Further, there are data indicating reduced mitochondrial respiration in tissue and cells from Black adults. Recent data from preclinical models and patients with hypertension suggest that depletion of SIRT3 leads to hyperacetylation (i.e., inactivation) of the mitochondrial antioxidant SOD2, which reduces endogenous antioxidant capacity, thus contributing to excessive oxidative stress and vascular dysfunction. Importantly, these findings have also been extended to PBMCs. However, the consideration of this SIRT3" SOD2 inactivation"excess mitochondrial ROS milieu has not been considered in the context of racial disparities in vascular dysfunction and BP regulation. MitoQ (Antipodean Pharmaceuticals) is a dietary supplement produced by covalently bonding ubiquinone, an endogenous mitochondrial antioxidant, and component of the electron transport chain, to a triphenylphosphonium cation to target mitochondria. Over 350 publications including multiple phase II trials have used MitoQ. Rodent findings exhibit that MitoQ accumulates in the vasculature to reduce both circulating and local (i.e., aorta homogenate) ROS. A prior human study that assigned older (60-79 yrs old) adults with impaired endothelial function to six weeks of oral MitoQ supplementation (20 mg/day) demonstrated a 42% improvement in endothelial function in a predominately White cohort. While MitoQ and SOD2 act through different mechanisms, both antioxidants act to reduce mitochondrial-derived oxidative stress. Thus, the investigators are seeking to leverage MitoQ which is commercially available, safe, and has a record of efficacy, to reduce mitochondrial ROS in Black adults, who the investigators hypothesize have reduced endogenous antioxidant activity via the SIRT3 SOD2 inactivation excess mitochondrial ROS milieu.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 45-75
* Have blood pressure no higher than 150/90 mmHg
* Have a BMI less than 40 Kg/m2 (otherwise healthy)
* Free from metabolic disease (diabetes or renal disease), pulmonary disorders (e.g., COPD & cystic fibrosis), and cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular)
* Free of any medical issues that prevent participants from exercising (i.e., cardiovascular issues, or muscle/joint issues including painful arthritis), giving blood (i.e., blood thinners), or allergies associated with MitoQ substances.

Exclusion Criteria:

* Known allergy to MitoQ
* High blood pressure - greater the 150/90 mmHg
* Low blood pressure - less than 90/50 mmHg
* History of cardiovascular disease
* History of cancer
* History of diabetes
* History of kidney disease
* Obesity (BMI > 40 kg/m2)
* Current pregnancy
* Nursing mothers
* Communication barriers

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Changes in flow-mediated dilation (FMD) | Changes from before and after 8 week supplementation and placebo
  Flow-mediated vasodilation will be assessed using continuous measures of brachial artery diameter and velocity via duplex Doppler ultrasound (Hitachi Arietta 70). The brachial artery will be imaged in the longitudinal plane proximal to the medial epicondyle using a high-frequency (6-12 MHz) linear-array probe. The ultrasound probe will be stabilized using a custom-built clamp. Shear rate (sec-1) will be calculated as [(blood flow velocity (cm*s-1) *4)/blood vessel diameter (mm)] The image will be recorded throughout a 60-s baseline, a 300-s ischemic stimulus (250 mmHg), and 180 seconds post deflation. FMD will be expressed as % dilation (final diameter-baseline diameter/baseline diameter x 100) and also normalized to the shear stimulus. Allometric scaling will be used if appropriate, including if there are baseline differences in artery diameter by race or condition.
Changes in pulse wave analysis (PWA) | Changes from before and after 8 week supplementation and placebo
  The investigators will use the SphygmoCor XCEL system to assess pulse wave analysis (PWA). A high-fidelity strain-gauge transducer is used to obtain the pressure waveform at the brachial pulse. PWA will be expressed as % (calculated as augmentation pressure divided by the pulse pressure).
Changes in pulse wave velocity (PWV) | Changes from before and after 8 week supplementation and placebo
  The investigators will use the SphygmoCor XCEL to assess pulse wave velocity (PWV). Distances from the carotid artery sampling site to the femoral artery (upper leg instrumented with a thigh cuff for oscillometric sphygmomanometry), and from the carotid artery to the suprasternal notch will be recorded. PWV will be expressed as cm/s
Changes in blood pressure reactivity | Changes from before and after 8 week supplementation and placebo
  The investigators will measure systolic and diastolic pressure using photoplethysmography at the finger. Systolic and diastolic blood pressure will be assessed at rest and during handgrip exercise. Blood pressure reactivity will be expressed as a change in pressure (mmHg) from baseline to a predetermined time during the stressor (e.g., minute one average and minute two average).
Changes in circulating reactive oxygen species | Changes from before and after 8 week supplementation and placebo
  The investigators will use electron paramagnetic resonance to measure reactive oxygen species (spectra units) in whole blood samples treated with a spin probe.
Changes in blood biomarkers of nitric oxide bioavailability | Changes from before and after 8 week supplementation and placebo
  The investigators will measure nitric oxide metabolites (nitrate and nitrite nanomolar concentration).

SECONDARY OUTCOMES:
Objective sleep duration | Baseline pre-intervention (14-days)
  Philips actiwatch spectrum will be used to quantify sleep duration. Participants will wear the watch units for 14 days. The investigators will assess actigraphy wear times with a sleep diary.
Objective sleep efficiency | Baseline pre-intervention (14-days)
  Philips actiwatch spectrum will be used to quantify sleep efficiency. Participants will wear the watch units for 14 days.
Subjective sleep quality | Baseline (pre-intervention)
  The investigators will administer the Pittsburgh Sleep Quality Index to assess perceived sleep quality reflective of the one-month period leading into the study. Each question is scored 0 to 3 starting with "Not during the past month", "Less than once a week", "Once or twice a week", and "Three or more times a week" Answers are cross-referenced between 7 domains for a total score to identify on paper if a person is a good sleeper or a poor sleeper. Higher scores are worse.
Subjective sleepiness | Baseline (pre-intervention)
  The investigators will administer the Epworth Sleepiness Scale (ESS), a questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Subjective sleep chronotype | Baseline (pre-intervention)
  The investigators will administer the Munich Chronotype Questionnaire which asks questions about work day and free day sleep schedules, work details, and lifestyle to provide data to aid in the understanding of how biological clocks work in social life. The Munich Chronotype Questionnaire categorizes each participant into one of seven chronotype groups, and utilizes data on participants' midsleep phase and sleep debt to survey what "type" of sleeper each person is.
Subjective insomnia | Baseline (pre-intervention)
  The investigators will administer the Insomnia Severity Index (which is a brief instrument that was designed to assess the severity of both nighttime and daytime components of insomnia. The questionnaire asks questions related to the last two weeks of sleep related to insomnia problems. There are 7 questions in total and the scale is 0 (none), 1 (mild), 2 (moderate), 3 (severe), and 4 (very severe). Higher scores are worse.
Subjective mood states | Baseline (pre-intervention)
  The investigators will administer the Profile of Mood States (POMS) which is a psychological rating scale used to assess transient, distinct mood states. The POMS measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment.
Subjective social status | Baseline (pre-intervention)
  The investigators will administer the MacArthur Scale of Subjective Social Status which is a pictorial representation that uses a symbolic ladder, developed to capture the common sense of social status based on usual socioeconomic status indicators. It has the additional advantage to allow comparisons between studies conducted in different populations.
Subjective childhood experiences | Baseline (pre-intervention)
  The investigators will administer the Philadelphia Adverse Childhood Experiences Survey (PHL ACEs) which measures childhood exposure to trauma. The PHL ACEs contains two subscales: the Conventional Adverse Childhood Experiences (Conventional ACEs) subscale and the Expanded Adverse Childhood Experiences (Expanded ACEs) subscale. There are 21 questions related to adverse childhood experiences. The scale is 1 (More than once), 2 (Once), and 3 (Never). A lower ACEs score is better.
Mental health - depression | Baseline (pre-intervention)
  The investigators will administer the Beck's Depression Inventory. The scale starts at 0 and ends at 3 for 21 questions related to depression.
Physical activity | Baseline pre-intervention (14-days)
  Participants will wear an ActiGraph GT3X accelerometer for fourteen days to objectively quantify steps per day
Habitual dietary intake | Baseline (pre-intervention)
  The investigators will instruct participants to complete a diet log for 5 days which will be operationalized with Nutrition Data System for Research (NDSR).
Subjective sleep apnea | Baseline (pre-intervention)
  The investigators will administer the Stop Bang Sleep Apnea Questionnaire which screens for obstructive sleep apnea (OSA) only, not central sleep apnea. The questionnaire consists of questions geared towards identifying if a person has sleep apnea (e.g., snoring, tiredness) and the scale is "Yes" or "No". A higher score is worse.
Subjective socioeconomic status | Baseline (pre-intervention)
  The investigators will administer the SES which measures participant responses coded and added to provide an index of childhood SES, adulthood SES, and lifetime SES (childhood + adulthood SES).

CONTACTS AND LOCATIONS:
Overall Officials: Austin T Robinson, PhD, Principal Investigator — Kinesiology Building
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate DMDA approvals
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after completion of the trial, indefinitely
Access Criteria: A formal plan identifying the intended use of the data and proper completion of a DMDA and MTA (if needed) with Auburn University and the study PI.

REFERENCES:
- [Background] Gane EJ, Weilert F, Orr DW, Keogh GF, Gibson M, Lockhart MM, Frampton CM, Taylor KM, Smith RA, Murphy MP. The mitochondria-targeted anti-oxidant mitoquinone decreases liver damage in a phase II study of hepatitis C patients. Liver Int. 2010 Aug;30(7):1019-26. doi: 10.1111/j.1478-3231.2010.02250.x. Epub 2010 May 18. PMID 20492507
- [Background] Snow BJ, Rolfe FL, Lockhart MM, Frampton CM, O'Sullivan JD, Fung V, Smith RA, Murphy MP, Taylor KM; Protect Study Group. A double-blind, placebo-controlled study to assess the mitochondria-targeted antioxidant MitoQ as a disease-modifying therapy in Parkinson's disease. Mov Disord. 2010 Aug 15;25(11):1670-4. doi: 10.1002/mds.23148. PMID 20568096
- [Background] Rossman MJ, Santos-Parker JR, Steward CAC, Bispham NZ, Cuevas LM, Rosenberg HL, Woodward KA, Chonchol M, Gioscia-Ryan RA, Murphy MP, Seals DR. Chronic Supplementation With a Mitochondrial Antioxidant (MitoQ) Improves Vascular Function in Healthy Older Adults. Hypertension. 2018 Jun;71(6):1056-1063. doi: 10.1161/HYPERTENSIONAHA.117.10787. Epub 2018 Apr 16. PMID 29661838
- [Background] Gioscia-Ryan RA, Battson ML, Cuevas LM, Eng JS, Murphy MP, Seals DR. Mitochondria-targeted antioxidant therapy with MitoQ ameliorates aortic stiffening in old mice. J Appl Physiol (1985). 2018 May 1;124(5):1194-1202. doi: 10.1152/japplphysiol.00670.2017. Epub 2017 Oct 26. PMID 29074712